CLINICAL TRIAL: NCT06174961
Title: The Effect of Exercise on Pharmacodynamics and Pharmacokinetics of a Single Dose of Unfractionated Heparin: A Randomized, Controlled, Cross-over Study
Brief Title: The Effect of Exercise on Pharmacodynamics and Pharmacokinetics of a Single Dose of Unfractionated Heparin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kristian Karstoft (Other)
Responsible Party: Sponsor-Investigator, Kristian Karstoft, Chief Physician, Principal Investigator, MD, PhD, DMSc, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-000150-20
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Blood Coagulation Disorder
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Unfractionated heparin + No exercise (Experimental): 15,000 units of unfractionated heparin will be administered in the thigh. No exercise will be performed afterwards.
  Interventions: Drug: Unfractionated heparin; Behavioral: No exercise
- Unfractionated heparin + Double-legged cycle ergometer exercise (Experimental): 15,000 units of unfractionated heparin will be administered in the thigh. Double-legged cycle ergometer exercise will be performed for 1 hour afterwards
  Interventions: Drug: Unfractionated heparin; Behavioral: Double-legged cycle ergometer exercise
- Unfractionated heparin + Single-legged ipsilateral cycle ergometer exercise (Experimental): 15,000 units of unfractionated heparin will be administered in the thigh. Single-legged cycle ergometer exercise in leg where unfractionated heparin injection is given will be performed for 1 hour afterwards
  Interventions: Drug: Unfractionated heparin; Behavioral: Single-legged cycle ergometer exercise, with unfractionated heparin injection in the exercising leg
- Unfractionated heparin + Single-legged contralateral cycle ergometer exercise (Experimental): 15,000 units of unfractionated heparin will be administered in the thigh. Single-legged cycle ergometer exercise in contralateral leg to where unfractionated heparin injection is given will be performed for 1 hour afterwards
  Interventions: Drug: Unfractionated heparin; Behavioral: Single-legged cycle ergometer exercise, with unfractionated heparin injection in the non-exercising leg

INTERVENTIONS:
Drug: Unfractionated heparin — 15,000 units of unfractionated heparin administered in the thigh
Behavioral: Double-legged cycle ergometer exercise — One hour of double-leg cycle ergometer exercise
  Arms: Unfractionated heparin + Double-legged cycle ergometer exercise
Behavioral: Single-legged cycle ergometer exercise, with unfractionated heparin injection in the exercising leg — One hour of single-leg cycle ergometer exercise, after unfractionated heparin injection in the ipsilateral leg
  Arms: Unfractionated heparin + Single-legged ipsilateral cycle ergometer exercise
Behavioral: Single-legged cycle ergometer exercise, with unfractionated heparin injection in the non-exercising leg — One hour of single-leg cycle ergometer exercise, after unfractionated heparin injection in the ipsilateral leg
  Arms: Unfractionated heparin + Single-legged contralateral cycle ergometer exercise
Behavioral: No exercise — No exercise
  Arms: Unfractionated heparin + No exercise

SUMMARY:
The aim of this project is to assess the influence of exercise on pharmacokinetics (PK) and pharmacodynamics (PD) of a single dose of subcutaneously (sc) administered unfractionated heparin (UFH). It is hypothesized that exercise will increase the systemic exposure (PK) and therefore the clinical effects (PD) of the sc administered UFH.

To assess this, healthy male volunteers will be included in a controlled, randomized, crossover study, where they, on four separate days, will have UFH injected sc in the thigh, followed by different exercise interventions (one per experimental day). Blood sampling, with the aim of assessing PK and PD will be performed during the following hours.

ELIGIBILITY:
Inclusion Criteria:

* Body weight 50 kg or more
* Body Mass Index 18.5-25 kg/m2
* Acceptance of not drinking alcohol for 24 hours before to 24 hours after dosing of study drug
* Acceptance of not performing physical activity for 24 hours before to 24 hours after dosing of study drug
* Signed informed consent form

Exclusion Criteria:

* History or sign of bleeding disorders
* History or sign of kidney disease
* History or sign of liver disease
* Average systolic blood pressure <100 mmHg or >140 mmHg and/or average diastolic blood pressure <60 mmHg or >90 mmHg (average of three measurements performed at screening).
* Daily pharmaceutical treatment
* Contraindication to increased levels of physical activity (10)
* Smoking or other regular use of any form of nicotine products during the study period and the previous 3 months.
* Current or prior participation (within 3 months before screening) in other clinical trials that might affect the results of this study (judged by the investigator).
* Previous treatment with heparins
* Low levels of anti-thrombin (P-antitrombin(enz.) <0,80 kIU/L)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Difference between interventions in change in incremental activated partial thromboplastin time (aPTT) | Peak aPTT for 1-8 hours after unfractionated heparin (UFH) injection

SECONDARY OUTCOMES:
Difference between interventions in change in incremental plasma heparin | Peak plasma heparin for 1-8 hours after UFH injection
Difference between interventions in mean incremental aPTT | 1-8 hours after UFH injection
Difference between interventions in mean incremental plasma heparin | 1-8 hours after UFH injection
Difference between interventions in change in aPTT | 4 hours after UFH injection
Difference between interventions in change in plasma heparin | 4 hours after UFH injection
Difference between interventions in mean incremental natriuretic peptides | 1-8 hours after UFH injection
Difference between interventions in mean incremental follistatin | 1-8 hours after UFH injection

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Karstoft, MD, DMSc, Principal Investigator — Bispebjerg-Frederiksberg Hospital, Department of Clinical Pharmacology
Locations (1):
- Bispebjerg-Frederiksberg Hospital, Department of Clinical Pharmacology, Copenhagen, Denmark